CLINICAL TRIAL: NCT02048566
Title: ImaCor II Effects of Hemodynamic Monitoring Using the ImaCor Single Use Transesophageal Echocardiography Probe in Critically Ill Patients - a Randomized Controlled Trial
Brief Title: Effects of Hemodynamic Monitoring Using the ImaCor Single Use Transesophageal Echocardiography Probe in Critically Ill Patients
Acronym: ImaCor II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: ImaCor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 174/13
Record Dates: First submitted 2014-01-21; First posted 2014-01-29 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Shock
Keywords: Echocardiography, Transesophageal; Monitoring, Physiologic; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- hTEEPM (Experimental): Group hTEE protocolled monitoring (hTEEPM) will receive echocardiography-guided hemodynamic management (hTEE) at the time of inclusion, at the time of occurrence of defined new organ system deterioration (see below) and/or at least every 4 hours during the first 72h after study inclusion or until one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Interventions: Device: ImaCor PM
- hTEESM (Experimental): Group hTEE standard monitoring (hTEESM) will receive echocardiography-guided hemodynamic management (hTEE) at the time of inclusion, follow-up assessment intervals are at the discretion of the treating physician for the first 72h after study inclusion. A follow up assessment is defined as any assessment that leads to significant changes in hemodynamic management in which case an hTEE assessment has to be performed. hTEE monitoring is discontinued if one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Interventions: Device: ImaCor SM
- ControlPM (Active Comparator): Group Control protocolized monitoring (ControlPM) will receive any hemodynamic monitoring of choice of the treating physician except ImaCor. Protocolized hemodynamic assessments will be performed at the time of inclusion, at the time of occurrence of defined new organ system deterioration or at least every 4 hours for the first 72h after study inclusion. Protocolized monitoring is discontinued if one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Interventions: Other: Control PM
- ControlSM (Active Comparator): Group Control standard monitoring (ControlSM) will receive any hemodynamic monitoring of choice of the treating physician except ImaCor. Protocolized hemodynamic assessments will be performed at the time of inclusion, follow-up measurement intervals are at the discretion of the treating physician for the first 72h after study inclusion. A follow up assessment is defined as any assessment that leads to significant changes in hemodynamic management. Data collection from standard monitoring is discontinued if one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Interventions: Other: Control SM

INTERVENTIONS:
Device: ImaCor PM — The ImaCor ClariTEE (hTEE) device is a transesophageal echocardiography system. It produces a single-plane two-dimensional image. The ImaCor probe is a 5.5 mm detachable probe; it can remain in situ for up to 72h and allows for reassessment of the patient's hemodynamic progress and the effect of selected interventions at any time. The probe is connected to a dedicated echocardiographic system which allows the for the recording of digital loops and performance of basic two-dimensional measurements. ImaCorPM subjects will receive echocardiography-guided hemodynamic management (hTEE) at the time of inclusion, at the time of occurrence of defined new organ system deterioration and/or at least every 4 hours during the first 72h after study inclusion or until one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Arms: hTEEPM
Device: ImaCor SM — The ImaCor ClariTEE (hTEE) device is a transesophageal echocardiography system. It produces a single-plane two-dimensional image. The ImaCor probe is a 5.5 mm detachable probe; it can remain in situ for up to 72h and allows for reassessment of the patient's hemodynamic progress and the effect of selected interventions at any time. The probe is connected to a dedicated echocardiographic system which allows the for the recording of digital loops and performance of basic two-dimensional measurements. ImaCorSM subjects will receive echocardiography-guided hemodynamic management (hTEE) at the time of inclusion, follow-up assessment intervals are at the discretion of the treating physician for the first 72h after study inclusion. hTEE monitoring is discontinued if one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Arms: hTEESM
Other: Control PM — Group Control protocolized monitoring (ControlPM) will receive any hemodynamic monitoring of choice of the treating physician except ImaCor. Protocolized hemodynamic assessments will be performed at the time of inclusion, at the time of occurrence of defined new organ system deterioration or at least every 4 hours for the first 72h after study inclusion. Protocolized monitoring is discontinued if one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Arms: ControlPM
Other: Control SM — Group Control standard monitoring (ControlSM) will receive any hemodynamic monitoring of choice of the treating physician except ImaCor. Protocolized hemodynamic assessments will be performed at the time of inclusion, follow-up measurement intervals are at the discretion of the treating physician for the first 72h. Data collection from standard monitoring is discontinued if one of the following events occurs: study primary endpoints reached, patient is extubated, withdrawal of active treatment.
  Arms: ControlSM

SUMMARY:
Hemodynamic management of critically ill patients is a constant challenge in the intensive care unit (ICU). Commonly used monitoring parameters to guide hemodynamic management generally consist of measurements of pressures (systemic and pulmonary artery pressures, cardiac filling pressures) and flow (cardiac output measurements using a thermodilution method). However, cardiac filling pressures and flow data have known limitations and might not accurately represent cardiac preload and contractility. Hemodynamic management of critically ill patients based on these parameters might therefore not be optimal and delay stabilisation of the patient, leading to negative outcomes and increased use of resources.

Visualization of the heart using echocardiography offers the advantage of direct measurement of cardiac volumes and systolic function. Echocardiography has been established as a tool to evaluate the causes of hemodynamic instability in ICU patients by the visualization of cardiac chambers, valves and pericardium and cardiac functional abnormalities. A repeated echocardiographic assessment could potentially provide useful additional information resulting in more rapid resolution of hemodynamic instability. Using conventional TTE and TEE, however, limits the feasibility of such an approach due to a lack of time and availability of appropriately trained staff.

In recently published studies the feasibility of hemodynamic monitoring and safety of hTEE was demonstrated. In the context of a prospective quality review assessment, the investigators showed that the echocardiographic examinations using hTEE were of sufficient quality in a majority of examined ICU patients and that the inter-rater reliability between the intensivists and a trained cardiologist was substantial. However, as of yet studies assessing the impact of hemodynamic monitoring by hTEE on relevant patient outcomes are not available. Given the associated costs for the hTEE device and the ultrasound probes and the additional resource requirements for training and application, the efficacy and efficiency of hTEE monitoring in comparison to standard monitoring should be established.

DETAILED DESCRIPTION:
Background

Hemodynamic management of critically ill patients is a constant challenge in the intensive care unit (ICU). Commonly used monitoring parameters to guide hemodynamic management generally consist of measurements of pressures (systemic and pulmonary artery pressures, cardiac filling pressures) and flow (cardiac output measurements using a thermodilution method). However, cardiac filling pressures and flow data have known limitations and might not accurately represent cardiac preload and contractility. To date, continuous or sequential recording of hemodynamic parameters is limited to pulse pressure variation measurement and indicator dilution techniques. The overall accuracy of these methods is not well established and comparisons of measurements of cardiac function parameters have been reported to trend differently in response to therapy and show limited interdevice agreement. Hemodynamic management of critically ill patients based on these parameters might therefore not be optimal and delay stabilisation of the patient, leading to negative outcomes and increased use of resources.

Visualization of the heart using echocardiography offers the advantage of direct measurement of cardiac volumes and systolic function. Echocardiography has been established as a tool to evaluate the causes of hemodynamic instability in ICU patients by the visualization of cardiac chambers, valves and pericardium and cardiac functional abnormalities. Transthoracic echocardiography (TTE) can be used as a first-line approach for a quick and focused examination to diagnose acute cor pulmonale, cardiac tamponade or major left ventricular systolic dysfunction. The training necessary to reliably perform such an abbreviated TTE use is substantial and the method is not readily available for every intensivist. Transesophageal echocardiography (TEE) can have a better diagnostic capability and is more reproducible than TTE. A minimum number of 31 TEE examinations has been reported to be required for intensivists to achieve competence in TEE driven hemodynamic evaluation of ventilated ICU patients. Additionally, repeatedly inserting the TEE probe as required for serial evaluation of a patients hemodynamic status is associated with a small but significant risk of injury to oral and esophageal structures. A repeated echocardiographic assessment could potentially provide useful additional information resulting in more rapid resolution of hemodynamic instability. Using conventional TTE and TEE, however, limits the feasibility of such an approach due to a lack of time and availability of appropriately trained staff.

In a recently published study the feasibility of hemodynamic monitoring and safety of hTEE was demonstrated in a group of ninety-four ventilated critically ill patients. In this study hTEE examinations were performed by four highly trained intensivist with extensive expertise in critically care echocardiography. The Department of Intensive Care Medicine Inselspital (KIM) has introduced hTEE in January 2012. The feasibility and quality of hemodynamic monitoring using hTEE by the department's intensivists was assessed in the context of a prospective quality review assessment. The study showed that the echocardiographic examinations using hTEE were of sufficient quality in a majority of examined ICU patients and that the inter-rater reliability between the intensivists and a trained cardiologist was substantial. However, as of yet studies assessing the impact of hemodynamic monitoring by hTEE on relevant patient outcomes are not available. Given the associated costs for the hTEE device and the ultrasound probes and the additional resource requirements for training and application, the efficacy and efficiency of hTEE monitoring in comparison to standard monitoring should be established.

The investigated device consists of a newly developed, commercially available transesophageal echocardiography system. The ImaCor ClariTEE technology (hTEE) device produces a single-plane two-dimensional image and has color Doppler capability (IMACOR, New-York NY, USA). The ImaCor probe is a 5.5 mm detachable probe; due to its small size it can remain in situ for up to 72h and therefore allows for reassessment of the patient's hemodynamic progress and the effect of selected interventions at any time. The probe has to be disposed after 72h for hygienic reasons. The probe is connected to a dedicated echocardiographic system which allows the recording of digital loops and performance of basic two-dimensional measurements of areas and distances. It provides a robust, but more rapid and user-friendly approach to monitoring hemodynamic status and cardiac function than conventional TTE/TEE.

Objective

The study hypothesis is that hemodynamic monitoring using hTEE of critically ill patients with hemodynamic compromise allows for an expedited reversal of circulatory impairment compared to standard ICU monitoring.

Primary Objective: To assess the impact of hemodynamic monitoring using the ImaCor ClariTEE technology on duration and amount of vasopressor use and time to reversal of shock in hemodynamically compromised patients in comparison to standard monitoring.

Secondary Objective: To assess the safety and tolerability of the ImaCor ClariTEE probe.

Methods

Subjects will be assigned to one of four groups stratified by method of hemodynamic monitoring (ImaCor vs control hemodynamic monitoring) and frequency of hemodynamic assessments (protocolized intervals PM vs standard monitoring intervals SM). In patients randomized to echocardiography-guided hemodynamic management (ImaCorPM and ImaCorSM) the ImaCor ClariTEE system will be installed at the time of study inclusion. An ICU consultant will assess the patients' hemodynamic condition based on the hTEE information (ImaCorPM and SM) and other available hemodynamic parameters (ControlPM and SM). Any changes in hemodynamic management are recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older AND
* Mechanical ventilation AND
* Systemic mean blood pressure < 60 mmHg (or < 80 mmHg if the patient has baseline hypertension) for more than 30 minutes despite adequate fluid resuscitation (minimum of 20 ml/kg crystalloids) OR
* Maintaining the systemic mean blood pressure > 60 mmHg requires any dose of vasopressors or inotropes AND at least one of the following:
* Capillary refilling time three seconds or longer
* Lactate >2 mmol/L
* Urine output <0.5 mL/kg for at least one hour
* Written informed consent

Exclusion Criteria

* Unrepaired tracheoesophageal fistula
* History of prior esophageal or gastric surgery precluding the use of TEE
* Esophageal obstruction or stricture
* Esophageal varices or diverticulum
* Esophageal or gastric perforation
* Gastric or esophageal bleeding
* Vascular ring, aortic arch anomaly with or without airway compromise
* Recent oropharyngeal surgery
* Severe coagulopathy (defined as thrombocyte count less than 30x10e9/l or INR > 3)
* Cervical spine injury or anomaly
* Elective ICU admission after elective surgery
* Use of cardiac assist devices
* Use of extra-corporeal membrane oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Time to resolution of hemodynamic instability as defined by systemic mean blood pressure > 60mmHg | At least 4 hours after discontinuation of vasopressors or inotropes

SECONDARY OUTCOMES:
Length of time with need for organ support (mechanical ventilation, renal-replacement therapy) | End of study, expected to be up to 24 weeks
Length of stay in the ICU | End of study, expected to be up to 24 weeks
Length of stay in the hospital | End of study, expected to be on average 1 year (or until death)
Signs of hypoperfusion or organ dysfunction (Capillary refill time, urinary output, blood lactate levels) | 72 hours
Use of conventional hemodynamic monitoring (PA catheter, CVP) | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tobias M Merz, PD Dr. med., Principal Investigator — Dep. of Intensive Care Medicine, Bern University Hospital; Jukka Takala, Prof. Dr. med., Study Chair — Dep. of Intensive Care Medicine, Bern University Hospital; Stephan M Jakob, Prof. Dr. med., Study Director — Dep. of Intensive Care Medicine, Bern University Hospital
Locations (1):
- Dep. of Intensive Care Medicine, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Vignon P, Mentec H, Terre S, Gastinne H, Gueret P, Lemaire F. Diagnostic accuracy and therapeutic impact of transthoracic and transesophageal echocardiography in mechanically ventilated patients in the ICU. Chest. 1994 Dec;106(6):1829-34. doi: 10.1378/chest.106.6.1829. PMID 7988209
- [Background] Jensen MB, Sloth E, Larsen KM, Schmidt MB. Transthoracic echocardiography for cardiopulmonary monitoring in intensive care. Eur J Anaesthesiol. 2004 Sep;21(9):700-7. doi: 10.1017/s0265021504009068. PMID 15595582
- [Background] Au SM, Vieillard-Baron A. Bedside echocardiography in critically ill patients: a true hemodynamic monitoring tool. J Clin Monit Comput. 2012 Oct;26(5):355-60. doi: 10.1007/s10877-012-9385-6. Epub 2012 Jul 27. PMID 22836724
- [Background] Vieillard-Baron A, Slama M, Mayo P, Charron C, Amiel JB, Esterez C, Leleu F, Repesse X, Vignon P. A pilot study on safety and clinical utility of a single-use 72-hour indwelling transesophageal echocardiography probe. Intensive Care Med. 2013 Apr;39(4):629-35. doi: 10.1007/s00134-012-2797-4. Epub 2013 Jan 4. PMID 23287876
- [Background] Cioccari L, Baur HR, Berger D, Wiegand J, Takala J, Merz TM. Hemodynamic assessment of critically ill patients using a miniaturized transesophageal echocardiography probe. Crit Care. 2013 Mar 27;17(3):R121. doi: 10.1186/cc12793. PMID 23786797
- [Derived] Merz TM, Cioccari L, Frey PM, Bloch A, Berger D, Zante B, Jakob SM, Takala J. Continual hemodynamic monitoring with a single-use transesophageal echocardiography probe in critically ill patients with shock: a randomized controlled clinical trial. Intensive Care Med. 2019 Aug;45(8):1093-1102. doi: 10.1007/s00134-019-05670-6. Epub 2019 Jul 4. PMID 31273416
- [Derived] Cioccari L, Zante B, Bloch A, Berger D, Limacher A, Jakob SM, Takala J, Merz TM. Effects of hemodynamic monitoring using a single-use transesophageal echocardiography probe in critically ill patients - study protocol for a randomized controlled trial. Trials. 2018 Jul 6;19(1):362. doi: 10.1186/s13063-018-2714-4. PMID 29980233

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT02048566/SAP_000.pdf